CLINICAL TRIAL: NCT01678677
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Non-typeable Haemophilus Influenzae (NTHi) Investigational Vaccine (GSK2838497A) in Current and Former Smokers
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of GSK Biologicals' Non-typeable Haemophilus Influenzae (NTHi) Investigational Vaccine (GSK2838497A) in Current and Former Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116647
Record Dates: First submitted 2012-08-23; First posted 2012-09-05 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders
Keywords: non-typeable Haemophilus influenzae; immunogenicity; reactogenicity; safety
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (10):
- Group A (Experimental): Subjects in this group will receive formulation 1 of NTHi vaccine.
  Interventions: Biological: NTHI vaccine GSK2838500A (formulation 1)
- Group B (Experimental): Subjects in this group will receive formulation 2 of NTHi vaccine.
  Interventions: Biological: NTHI vaccine GSK2838501A (formulation 2)
- Group C (Experimental): Subjects in this group will receive formulation 3 of NTHi vaccine.
  Interventions: Biological: NTHI vaccine GSK2838502A (formulation 3)
- Group D (Experimental): Subjects in this group will receive formulation 4 of NTHi vaccine.
  Interventions: Biological: NTHI vaccine GSK2838503A (formulation 4)
- Group E (Experimental): Subjects in this group will receive formulation 5 of NTHi vaccine and a placebo.
  Interventions: Biological: NTHI vaccine GSK2838504A (formulation 5)
- Group F (Experimental): Subjects in this group will receive formulation 6 of NTHi vaccine and a placebo.
  Interventions: Biological: NTHI vaccine GSK2838505A (formulation 6)
- Group G (Experimental): Subjects in this group will receive formulation 7 of NTHi vaccine and a placebo.
  Interventions: Biological: NTHI vaccine GSK2838508A (formulation 7)
- Group H (Experimental): Subjects in this group will receive formulation 8 of NTHi vaccine and a placebo.
  Interventions: Biological: NTHI vaccine GSK2838509A (formulation 8)
- Group Placebo 1 (Placebo Comparator): Subjects in this group will receive placebo.
  Interventions: Drug: Placebo comparator
- Group Placebo 2 (Placebo Comparator): Subjects in this group will receive placebo.
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Biological: NTHI vaccine GSK2838500A (formulation 1) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group A
Biological: NTHI vaccine GSK2838501A (formulation 2) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group B
Biological: NTHI vaccine GSK2838502A (formulation 3) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group C
Biological: NTHI vaccine GSK2838503A (formulation 4) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group D
Biological: NTHI vaccine GSK2838504A (formulation 5) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group E
Biological: NTHI vaccine GSK2838505A (formulation 6) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group F
Biological: NTHI vaccine GSK2838508A (formulation 7) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group G
Biological: NTHI vaccine GSK2838509A (formulation 8) — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group H
Drug: Placebo comparator — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Arms: Group Placebo 1; Group Placebo 2

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of 8 different formulations of investigational NTHI vaccine in current and former smokers, 50-70 years of age.

DETAILED DESCRIPTION:
This Protocol Posting has been updated following Protocol Amendment 1, dated 10 October 2012, leading to a change in an inclusion criterion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 50 and 70 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Subjects without medical history, clinical finding or laboratory finding which in the opinion of the investigator could pose a safety concern or interfere with the protocol.
* Current or former smokers.
* A smoking history of at least 10 pack-years.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine, with the exception of any influenza vaccine which may be administered ≥ 15 days preceding or following any study vaccine dose.
* Previous vaccination with any vaccine containing NTHi-antigens.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of or current autoimmune disease.
* Post-bronchodilator Forced Expiratory Volume in 1 second (FEV1) < 80% of predicted normal value.
* Diagnosed with a respiratory disorder. Please note that subjects with mild pulmonary obstruction can be enrolled.
* Laboratory evidence of clinically significant haematological abnormalities at Screening.
* Acute disease and/or fever at the time of enrolment.
* Current alcoholism and/or drug abuse.
* Has significant disease, in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.
* History of or current condition preventing intramuscular injection as bleeding or coagulation disorder.
* Has contraindication for spirometry testing.
* Malignancies within previous 5 years and lymphoproliferative disorders.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any other condition that the investigator judges may interfere with study findings.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2014-01-30 (Actual); Study Completion 2014-01-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of each solicited local and general adverse event (AE), in all subjects, in all groups. | During a 7-day follow-up period (from day 0 to day 6) after each vaccination.
Occurrence of any unsolicited AE, in all subjects, in all groups. | During a 30-day follow-up period (from day 0 to day 29) after each vaccination.
Occurrence of haematological and biochemical laboratory abnormalities, in all subjects, in all groups. | Prior to each vaccination.
Occurrence of haematological and biochemical laboratory abnormalities, in all subjects, in all groups. | 7 days after each vaccination.
Occurrence of haematological and biochemical laboratory abnormalities, in all subjects, in all groups. | At study conclusion (Day 420).
Occurrence of any serious adverse event (SAE), in all subjects, in all groups. | From first vaccination (Day 0) to study conclusion (Day 420).
Occurrence of any potential immune-mediated disease (pIMD) in all subjects, in all groups. | From first vaccination (Day 0) to study conclusion (Day 420).

SECONDARY OUTCOMES:
Humoral immune response to the components of the NTHi vaccine formulations, in all subjects, in all groups, in terms of antibody concentrations. | Prior to each vaccination, 30 days after each vaccination, and at study conclusion (Day 420).
Cell-mediated immune (CMI) responses to components of the NTHi vaccine formulations, in a sub-cohort of subjects, in all groups. | Prior to each vaccination, 30 days after each vaccination, and at study conclusion (Day 420).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Wilrijk

REFERENCES:
- See also: Results for study 116647 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/116647?search=study&b%22b''%22#rs